CLINICAL TRIAL: NCT05647772
Title: Reach and Scalability of Digital Therapeutics for Childhood Behavior Problems
Brief Title: Digital Therapeutics for Behavior Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Oliver Lindhiem, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY22030138; R01HD106930 (NIH)
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Problem Behavior; Child Behavior
Keywords: Oppositional Defiant Disorder (ODD); Conduct Disorder (CD); Childhood Behavioral Disorders; Mobile Health
MeSH Terms: conditions — Problem Behavior; Child Behavior; Oppositional Defiant Disorder; Conduct Disorder | interventions — Doulas

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial. The investigators will use stratified randomization to ensure that the groups are equivalent on key clinical features. Randomization will take place after completion of the initial baseline assessment. Parents of children (ages 5-8) with disruptive behaviors (N = 324 subjects) will be randomly assigned to Group 1 (standalone app; n = 108), Group 2 (coach-assisted app; n = 108), or Group 3 (control app; n = 108).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Standalone App (Experimental): Standalone parenting app called UseIt!
  Interventions: Behavioral: UseIt! App
- Group 2: App plus Coach (Experimental): Standalone parenting app called UseIt! plus a coach.
  Interventions: Behavioral: UseIt! App; Behavioral: Coach
- Group 3: Control App (Active Comparator): Control condition: mindfulness app called SmilingMind.
  Interventions: Behavioral: SmilingMind App

INTERVENTIONS:
Behavioral: UseIt! App — The UseIt! app is a parenting app with evidence-based parent management content. The app runs on both Android and iOS devices. It includes a digital library of parent management skills, a trouble-shooting guide, a behavior diary, a point counter, and a skills-alarm.
  Arms: Group 1: Standalone App; Group 2: App plus Coach
Behavioral: Coach — The coach is be a bachelor's level paraprofessional with a degree in psychology or an allied discipline (e.g., social work) who provides support to parents. The coach will provide motivation and accountability but will not provide therapeutic/clinical support. The primary goal of the coach is to increase participant engagement with the UseIt! mHealth system.
  Arms: Group 2: App plus Coach
Behavioral: SmilingMind App — The control app is a mindfulness app called SmilingMind. It is available for both Android and iOS devices.
  Arms: Group 3: Control App

SUMMARY:
In this project, the investigators aim to test the effectiveness of a mobile health (mHealth) system as a standalone versus coach-assisted intervention with the goal of achieving reach and scalability. Parents of children (ages 5-8) with disruptive behaviors (N = 324 subjects) will be randomly assigned to Group 1 (standalone app), Group 2 (coach-assisted app), or Group 3 (control app).

DETAILED DESCRIPTION:
In this project, the investigators aim to test the effectiveness of a mobile health (mHealth) system as a standalone versus coach-assisted intervention with the goal of achieving reach and scalability. Aim 1 is to evaluate the effectiveness of the UseIt! mHealth system as both a standalone and coach-assisted intervention compared to a control app condition. Aim 2 is to assess target (parent management training/cognitive behavioral therapy skill acquisition and use) engagement and validation. Aim 3 is to evaluate the effectiveness of the components of the UseIt! mHealth system. The investigators plan to recruit an anticipated total of 324 families for the study. Families will be randomly assigned to Group 1 (standalone app), Group 2 (coach-assisted), or Group 3 (control app condition). Parents will use the app for four months before the administration of the post-treatment assessment. Parents will be trained to use the UseIt! mHealth system over the phone. The coach for the Group 2 condition will be a bachelor's level paraprofessional with a degree in psychology or an allied discipline (e.g., social work) who will provide support to parents. The system is very user friendly and families can be trained in approximately 30 minutes. Assessments will take place at Baseline, Post (4 months from baseline), and 6-month follow-up. All assessments will be conducted online (Qualtrics survey links sent via email by research staff) and take approximately 1 hour to complete.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 5-8 years
* Above the 90th percentile for Oppositional Defiant Disorder (ODD) and/or conduct disorders (CD) on the Vanderbilt Assessment Scale
* Residence with at least one parent/guardian at least 80% of the time
* Parent/legal guardian consent for participation
* Parent/guardian must have a smartphone device with daily internet access

Exclusion Criteria:

* A known preexisting behavioral or mental health diagnosis requiring alternative treatment (bipolar disorder, major depression, pervasive developmental disorder)
* Currently in treatment for childhood disruptive behavior

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Effective Parenting Test (KEPT) | Post assessment (4 months after baseline).
  Average scores from the Knowledge of Effective Parenting Test (KEPT). This is a 21-item scale, with higher scores indicating better outcomes.
Knowledge of Effective Parenting Test (KEPT) | 6-month follow-up (10 months after baseline).
  Average scores from the Knowledge of Effective Parenting Test (KEPT). This is a 21-item scale, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Parenting Skill Use Diary (PSUD) | Post assessment (4 months after baseline).
  Average scores from the Parenting Skill Use Diary (PSUD). This is a proportion score (range 0 to 1), with higher scores indicating better outcomes.
Parenting Skill Use Diary (PSUD) | 6-month follow-up (10 months after baseline).
  Average scores from the Parenting Skill Use Diary (PSUD). This is a proportion score (range 0 to 1), with higher scores indicating better outcomes.
Oppositional Defiant Disorder Subscale of the Vanderbilt Assessment | Post assessment (4 months after baseline).
  Average scores from the Oppositional Defiant Disorder Subscale of the Vanderbilt Assessment. Scores range from 0 to 24, with higher scores indicating worse outcomes.
Oppositional Defiant Disorder Subscale of the Vanderbilt Assessment | 6-month follow-up (10 months after baseline).
  Average scores from the Oppositional Defiant Disorder Subscale of the Vanderbilt Assessment. Scores range from 0 to 24, with higher scores indicating worse outcomes.
Conduct Disorder Subscale of the Vanderbilt Assessment | Post assessment (4 months after baseline).
  Average scores from the Conduct Disorder Subscale of the Vanderbilt Assessment. Scores range from 0 to 42, with higher scores indicating worse outcomes.
Conduct Disorder Subscale of the Vanderbilt Assessment | 6-month follow-up (10 months after baseline).
  Average scores from the Conduct Disorder Subscale of the Vanderbilt Assessment. Scores range from 0 to 42, with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Lindhiem, PhD, Principal Investigator — University of Pittsburgh, Department of Psychiatry
Locations (1):
- Bellefield Towers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected for this project will be made available to other researchers for future data mining, following publication of primary findings at the conclusion of the study. The investigators will share data with other investigators within and outside the University of Pittsburgh upon submission of a standardized written request. All data sharing will follow the guidelines and rules of the NIH and our IRB. Data (both raw data and summary scores) will be shared electronically (secure digital file) as de-identified data.
Supporting Information: Study Protocol
Time Frame: Following publication of primary findings at the conclusion of the study.
Access Criteria: To gain access, anyone not part of the original research protocol will submit a Data Analysis Request Form which requires elucidation of hypotheses to be tested and specific data requested. This form requires information about the investigator, including institutional affiliation, resume, proposed research, and conflict of interest statement. The investigator must document completion of the University of Pittsburgh Certification Program in Research Practice Fundamentals or a comparable training program at their own institution. Investigators outside the University of Pittsburgh must also complete a Data Use and Confidentiality Agreement before release of data to them.

REFERENCES:
- [Derived] Lindhiem O, Tomlinson CS, Kolko DJ, Silk JS, Hafeman D, Wallace M, Setiawan IMA, Parmanto B. Novel Smartphone App and Supportive Accountability for the Treatment of Childhood Disruptive Behavior Problems: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 11;14:e67051. doi: 10.2196/67051. PMID 40068698